CLINICAL TRIAL: NCT00037206
Title: An Open Label Non-Comparative Study of the Safety and Efficacy of Intravenous Anidulafungin Plus AmBisome® [(Amphotericin B) Liposome for Injection] as a Treatment for Invasive Aspergillosis.
Brief Title: A Safety & Effectiveness Study of Intravenous Anidulafungin With AmBisome® for Treatment of Invasive Aspergillosis (IA).
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Vicuron Pharmaceuticals (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VER002-7; A8851001
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Aspergillosis
Keywords: Invasive Aspergillosis
MeSH Terms: conditions — Aspergillosis | interventions — Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin, VER002

SUMMARY:
The combination of Anidulafungin plus AmBisome® may offer an improved outcome for patients treated for Invasive Aspergillosis (IA). The purpose of this study is to determine the safety and the clinical and microbiological effectiveness of anidulafungin plus AmBisome® in treated patients located in the United States, Europe, and South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite IA outside the pulmonary system or definite or probable pulmonary IA
* Life expectancy: greater than 72 hours

Exclusion Criteria:

* Pregnant female
* Hypersensitivity to anidulafungin or echinocandin therapy
* Hypersensitivity to Tween 80 (polysorbate 80) or tartaric acid
* Hypersensitivity to amphotericin B deoxycholate or any other constituents of AmBisome unless, in the opinion of the investigator, the benefit of therapy outweighs the risk.
* Aspergilloma-in the absence of invasive disease
* Abnormal blood chemistries:

Bilirubin > 3 times the upper limit of normal; AST (aspartate aminotransferase) or ALT (alanine aminotransferase)> 5 times the upper limit of normal

* Greater than five days of therapeutic doses of systemic therapy for the current Aspergillus-associated condition or a cumulative dose of more than 5 mg/Kg of amphotericin, more than 25 mg/Kg of a lipid formulation of amphotericin, or more than 2g of itraconazole for the current condition. Prophylactic use of azoles or amphotericin is acceptable.
* Less than 4 weeks since prior participation in an investigational drug or device study, with the exception of cytotoxic, antiretroviral agents and therapies for AIDS-related opportunistic infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-05; Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Versicor, Inc., King of Prussia, Pennsylvania, United States